CLINICAL TRIAL: NCT00004920
Title: Phase III Study of Tomudex and Cisplatin Versus Cisplatin in Malignant Pleural Mesothelioma
Brief Title: Cisplatin With or Without Raltitrexed in Treating Patients With Malignant Mesothelioma of the Pleura
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-08983; EORTC-08983
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; raltitrexed

INTERVENTIONS:
Drug: cisplatin
Drug: raltitrexed

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether receiving cisplatin with raltitrexed is more effective than cisplatin alone for malignant mesothelioma.

PURPOSE: Randomized phase III trial to compare the effectiveness of cisplatin with or without raltitrexed in treating patients who have malignant mesothelioma of the pleura.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival in patients with malignant pleural mesothelioma treated with raltitrexed with or without cisplatin.
* Assess toxicity, progression free survival, and quality of life with these treatment regimens in these patients.
* Evaluate objective response and duration of response to these treatment regimens in patients with measurable disease.

OUTLINE: This is a randomized, open, multicenter study. Patients are stratified according to performance status (0 vs 1-2) and WBC count (less than 8,300/mm3 vs 8,300/mm3 or more). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive cisplatin IV over 1-2 hours on day 1.
* Arm II: Patients receive raltitrexed IV over 15 minutes followed by cisplatin IV over 1-2 hours on day 1.

Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before study, prior to each course, after the last course, and then every 6 weeks for 1 year.

Patients are followed every 6 weeks until death.

PROJECTED ACCRUAL: A total of 240 patients will be accrued for this study over 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant pleural mesothelioma
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ZUBROD, ECOG, WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 10.0 g/dL
* WBC at least 4,000/mm^3
* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.46 mg/dL
* Albumin at least 3.0 g/dL
* ALAT/ASAT less than 2.5 times upper limit of normal (ULN) (less than 5 times ULN if liver involvement)

Renal:

* Creatinine less than 1.69 mg/dL
* Creatinine clearance at least 65 mL/min

Cardiovascular:

* Not specified

Pulmonary:

* Not specified

Other:

* No other prior or concurrent malignancies within past 5 years except adequately treated carcinoma in situ of the cervix or basal or squamous cell carcinoma of the skin
* No prior malignant melanoma, hypernephroma or breast carcinoma
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* No uncontrolled infections
* No psychological, familial, sociological, or geographical condition that precludes study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy before first disease progression

Chemotherapy:

* No prior systemic or intracavitary cytotoxic chemotherapy
* No other prior or concurrent chemotherapy before first disease progression
* No prior or concurrent pleurodesis with cytotoxic drugs (e.g., bleomycin)

Endocrine therapy:

* No concurrent hormonal therapy except corticosteroids before first disease progression

Radiotherapy:

* At least 4 weeks since prior radiotherapy to target lesion and progression observed
* Concurrent palliative radiotherapy to painful lesions allowed only if target lesion outside of irradiated field

Surgery:

* Prior surgery allowed if followed by disease progression

Other:

* At least 1 month since prior investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 1999-11; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan P. Van Meerbeeck, MD, PhD, Study Chair — University Medical Center Rotterdam at Erasmus Medical Center
Locations (26):
- U.Z. Gasthuisberg, Leuven, Belgium
- Canada (6):
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- National Cancer Institute of Egypt, Cairo, Egypt
- France (3):
  - Assistance Publique Hopitaux de Marseille Hopitaux Sud, Marseille
  - Hopital de la Conception, Marseille
  - Hopital Charles Nicolle, Rouen
- Thoraxklinik Rohrbach, Heidelberg, Germany
- Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova), Italy
- Netherlands (4):
  - University Medical Center Nijmegen, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Erasmus Medical Center, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - Regional Lung Diseases Hospital, Poznan
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - St. Gallen, Sankt Gallen
- United Kingdom (3):
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Weston Park Hospital, Sheffield, England
  - Western General Hospital, Edinburgh, Scotland

REFERENCES:
- [Background] Francart J, Legrand C, Sylvester R, Van Glabbeke M, van Meerbeeck JP, Robert A. Progression-free survival rate as primary end point for phase II cancer clinical trials: application to mesothelioma--The EORTC Lung Cancer Group. J Clin Oncol. 2006 Jul 1;24(19):3007-12. doi: 10.1200/JCO.2005.05.1359. PMID 16809726
- [Result] Bottomley A, Coens C, Efficace F, Gaafar R, Manegold C, Burgers S, Vincent M, Legrand C, van Meerbeeck JP; EORTC-NCIC. Symptoms and patient-reported well-being: do they predict survival in malignant pleural mesothelioma? A prognostic factor analysis of EORTC-NCIC 08983: randomized phase III study of cisplatin with or without raltitrexed in patients with malignant pleural mesothelioma. J Clin Oncol. 2007 Dec 20;25(36):5770-6. doi: 10.1200/JCO.2007.12.5294. PMID 18089874
- [Result] Bottomley A, Gaafar R, Manegold C, Burgers S, Coens C, Legrand C, Vincent M, Giaccone G, Van Meerbeeck J; EORTC Lung-Cancer Group; National Cancer Institute, Canada. Short-term treatment-related symptoms and quality of life: results from an international randomized phase III study of cisplatin with or without raltitrexed in patients with malignant pleural mesothelioma: an EORTC Lung-Cancer Group and National Cancer Institute, Canada, Intergroup Study. J Clin Oncol. 2006 Mar 20;24(9):1435-42. doi: 10.1200/JCO.2005.03.3027. Epub 2006 Jan 30. PMID 16446322
- [Result] van Meerbeeck JP, Gaafar R, Manegold C, Van Klaveren RJ, Van Marck EA, Vincent M, Legrand C, Bottomley A, Debruyne C, Giaccone G; European Organisation for Research and Treatment of Cancer Lung Cancer Group; National Cancer Institute of Canada. Randomized phase III study of cisplatin with or without raltitrexed in patients with malignant pleural mesothelioma: an intergroup study of the European Organisation for Research and Treatment of Cancer Lung Cancer Group and the National Cancer Institute of Canada. J Clin Oncol. 2005 Oct 1;23(28):6881-9. doi: 10.1200/JCO.20005.14.589. PMID 16192580
- [Result] Van Meerbeeck JP, Manegold C, Gaafar R, et al.: A randomized phase III study of cisplatin with or without raltitrexed in patients (pts) with malignant pleural mesothelioma (MPM): an intergroup study of the EORTC Lung Cancer Group and NCIC. [Abstract] J Clin Oncol 22 (Suppl 14): A-7021, 622s, 2004.